CLINICAL TRIAL: NCT00182962
Title: Geriatric Resources for Assessment and Care of Elders
Brief Title: GRACE: Geriatric Resources for Assessment and Care of Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Nina Mason Pulliam Charitable Trust (Unknown); Wishard Health Services (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AG0042; R01AG020175 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-11-20 (Estimated); Status verified 2006-11

CONDITIONS: Functional Decline; Aging
Keywords: Activities of Daily Living; Low-income; geriatric medicine; computer assisted patient care
MeSH Terms: interventions — Restraint, Physical

INTERVENTIONS:
Behavioral: Geriatric Resources for Assessment & Care of Elders (GRACE)

SUMMARY:
The purpose of this study is to test the effectiveness of a collaborative model of team care as compared to usual care in improving functional outcomes among community-dwelling low-income older adults.

DETAILED DESCRIPTION:
This collaborative model of care, Geriatric Resources for Assessment and Care of Elders (GRACE), involves a geriatric nurse practitioner and a geriatric social worker caring for the vulnerable older adult in collaboration with the patient's primary care physician to improve coordination and quality of care. The specific components of GRACE mirror those recommended in recent reviews: a) specific targeting of elders at risk; b) availability of collaborative expertise in geriatrics; c) integration of the program into primary care; d) coordination of care across all sites of care; e) integration of data systems that support physician's practice and facilitate monitoring of pertinent clinical parameters; and f) institutionally endorsed clinical practice guidelines. To our knowledge, there are no prior studies investigating the effectiveness of such a comprehensive approach among vulnerable older adults.

We are hypothesizing that, compared to usual care, patients enrolled in the intervention will have:

1. greater independence in activities of daily living over 2 years of follow-up;
2. better health status scores as assessed by the HEDIS® 2000 Health Outcomes Survey
3. fewer nursing home days over 2 years of follow-up; and
4. fewer hospitalizations over the 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* Annual income less than 200% of the federal poverty level
* Have had one or more primary care visits in the past 12 months
* Reside in the community (non-institutionalized)

Exclusion Criteria:

* Non-English speaking
* No regular access to a telephone
* Currently undergoing kidney dialysis treatments
* Residing with a patient already participating in the GRACE clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1270
Dates: Start 2002-03; Study Completion 2006-10

PRIMARY OUTCOMES:
Functional status
health status
hospitalization and nursing home placement

SECONDARY OUTCOMES:
Patient satisfaction and quality of care

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Counsell, MD, Principal Investigator — Indiana University Geriatrics Program, Indiana University Center for Aging Research, Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Bernabei R, Landi F, Gambassi G, Sgadari A, Zuccala G, Mor V, Rubenstein LZ, Carbonin P. Randomised trial of impact of model of integrated care and case management for older people living in the community. BMJ. 1998 May 2;316(7141):1348-51. doi: 10.1136/bmj.316.7141.1348. PMID 9563983
- [Background] Callahan CM, Stump TE, Stroupe KT, Tierney WM. Cost of health care for a community of older adults in an urban academic healthcare system. J Am Geriatr Soc. 1998 Nov;46(11):1371-7. doi: 10.1111/j.1532-5415.1998.tb06003.x. PMID 9809758
- [Background] Counsell SR, Holder CM, Liebenauer LL, Palmer RM, Fortinsky RH, Kresevic DM, Quinn LM, Allen KR, Covinsky KE, Landefeld CS. Effects of a multicomponent intervention on functional outcomes and process of care in hospitalized older patients: a randomized controlled trial of Acute Care for Elders (ACE) in a community hospital. J Am Geriatr Soc. 2000 Dec;48(12):1572-81. doi: 10.1111/j.1532-5415.2000.tb03866.x. PMID 11129745
- [Background] Stuck AE, Minder CE, Peter-Wuest I, Gillmann G, Egli C, Kesselring A, Leu RE, Beck JC. A randomized trial of in-home visits for disability prevention in community-dwelling older people at low and high risk for nursing home admission. Arch Intern Med. 2000 Apr 10;160(7):977-86. doi: 10.1001/archinte.160.7.977. PMID 10761963
- [Background] Chen A, Brown R, Archibald N, Aliotta S, Fox PD. Best practice in coordinated care. Health Care Financing Administration. 2000. Contract No. HCFA 500-95-0048 (04).
- [Result] Counsell SR, Callahan CM, Buttar AB, Clark DO, Frank KI. Geriatric Resources for Assessment and Care of Elders (GRACE): a new model of primary care for low-income seniors. J Am Geriatr Soc. 2006 Jul;54(7):1136-41. doi: 10.1111/j.1532-5415.2006.00791.x. PMID 16866688
- [Result] Clark DO, Callahan CM, Counsell SR. Reliability and validity of a steadiness score. J Am Geriatr Soc. 2005 Sep;53(9):1582-6. doi: 10.1111/j.1532-5415.2005.53485.x. PMID 16137291
- [Derived] Counsell SR, Callahan CM, Tu W, Stump TE, Arling GW. Cost analysis of the Geriatric Resources for Assessment and Care of Elders care management intervention. J Am Geriatr Soc. 2009 Aug;57(8):1420-6. doi: 10.1111/j.1532-5415.2009.02383.x. PMID 19691149
- [Derived] Counsell SR, Callahan CM, Clark DO, Tu W, Buttar AB, Stump TE, Ricketts GD. Geriatric care management for low-income seniors: a randomized controlled trial. JAMA. 2007 Dec 12;298(22):2623-33. doi: 10.1001/jama.298.22.2623. PMID 18073358